CLINICAL TRIAL: NCT02329574
Title: Prediction of Persistent Post-Mastectomy Pain
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kristin Schreiber, Faculty, Department of Anesthesiology, Brigham and Women's Hospital
Other Study IDs: 2013P002202
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic pain is devastating both to individuals and society. In an aging population, surgery is an increasing cause of chronic pain, with rates of persistent post-operative pain ranging from 10-65%.In particular, Persistent Post-Mastectomy Pain (PPMP) occurs in roughly one third of women who have had mastectomy. The occurrence of PPMP does not seem to be strongly determined by the type of surgery, chemotherapy, and radiation treatment, suggesting that individual person-specific factors may play a more important role. In fact, recent studies indicate that individual differences in pain sensitivity (psychophysics) are more closely associated with PPMP than surgical/medical variables. Specifically, sensory testing revealed that women who developed PPMP had lower pressure pain thresholds and greater temporal summation of pain stimuli than women who did not develop this chronic pain condition. Moreover, psychosocial factors such as anxiety, depression, catastrophizing, and somatization were more prominent in women with PPMP. These preliminary, retrospective studies suggest that individual psychophysical and psychosocial characteristics could be important risk factors for PPMP. Accordingly, the aim of this study is to comprehensively and prospectively study women having mastectomy surgery, to determine the relationship between pre-operative psychophysical and psychosocial factors and the development of PPMP. Using these data, a prediction model for PPMP will be developed, thus allowing a preoperative calculation of a "PPMP risk score" for any patient facing mastectomy.

DETAILED DESCRIPTION:
This study is a prospective observational study which phenotypes individuals' baseline pain, psychosocial and psychophysical characteristics, then measures perioperative and long-term changes to examine the relationship of psychophysical and psychosocial processing to persistent post-mastectomy pain development .

Preoperative Psychophysical assessment:

Pressure pain testing methods: After giving informed consent, the PI or a fully trained member of the research staff will administer a brief QST session. Pressure pain threshold and tolerance will be assessed using a digital pressure algometer (Wagner FDX, Greenwich, CT, USA) with a flat round transducer, probe area 0.785 cm2. Testing sites will be bilateral on the dorsal aspect of the proximal forearm (extremity site) and over the trapezius muscle at the upper back (truncal site). For pressure threshold determination, pressure is increased at a steady rate of approximately 1 kg/second until subject indicates that the pressure is first perceived as painful. Pressure pain tolerance will be determined by instructing patients to indicate the pressure at which the pain was no longer tolerable. Two trials will be performed at each site.

Temporal Summation testing methods: Mechanical pinprick pain will be assessed using standardized weighted pinprick applicators similar to those described by Rolke et al99 of two designated forces (256mN and 512mN) which result in a painful sensation in most subjects.1-2,100 First, a single stimulation of the lower force pinprick will be applied to the dorsal aspect of the index finger between the first and second interphalangeal joints of the each hand while resting palm down on the armrest, and then rated by the subject on a scale of 0-10. Next, after a break of at least 10 seconds, a train of 10 stimuli will be applied at the same premarked spot, at a rate of 1 stimulation/second. The subject will rate pain on a scale of 0-10 after the first, fifth and tenth stimulus, then rate any ongoing pain 15 and 30 seconds after cessation of the last stimulus. The same procedure will be repeated using the higher force pinprick on the third finger of the each hand. Subjects will undergo two trials at each force, with a break of at least one minute between trials.

Psychosocial Assessment: Preoperative demographic, medical, psychosocial and pain questionnaires will be completed by the patient during their preoperative office visit. Questionnaires assessing psychosocial factors are chosen based upon previous association with PPMP, strong psychometric validation characteristics, and brevity. The Pain Catastrophizing Scale (PCS), which has been validated in pain patients and controls, will be used to measure catastrophic thinking associated with pain. Depressive symptoms, anxiety and sleep disturbance will be assessed using short-form instruments from the NIH roadmap initiative, Patient Reported Outcome Measurement Information System (PROMIS), which have been extensively validated in studies comparing results with established scales, and have been calibrated on over 20,000 persons. The Brief Symptom Index 18-Somatization Scale, also previously validated in chronic pain patients,107 will be used to measure somatization.

Pain assessment: The primary pain outcome measure will be Pain Burden Index as measured by the Breast Cancer Pain Questionnaire (BCPQ), which was originally developed by Gartner et al and used in over 600 patients in our previous studies. The BCPQ includes assessment of average pain, pain frequency (how many days/week), and pain location (breast, arm, side, axilla), from which an Pain Burden Index (PBI) can be calculated. The BCPQ also includes questions about other body pain, seeking medical help for pain, and painkiller use. We will also use the Brief Pain Inventory (BPI), a well-validated general measure of pain and disability worst pain, least pain, and interference. We will supplement this with questions assessing pain with and without movement. We will assess for neuropathic character of pain using the Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS).1 The Pain Coping Questionnaire will be administered to prospectively assay for effective coping strategies used by patients.

Medical, Anesthetic and Surgical Assessment: Medical variables, including patient's functional status, will be assessed at the preoperative visit. Using the Weiner preoperative evaluation center email alert system, the hands-on anesthetist and/or anesthesiologist will be contacted to inform them on the patient's participation in the study. In order to assess and adjust for potential impact of anesthetic technique or pharmacological agents on PPMP, the following data will be collected on the day of surgery: Primary anesthetic method (volatile agent vs. IV propofol vs. regional/paravertebral), amount and type of local anesthetic administered, and amount of opioids used (the latter expressed as morphine equivalent units/hr). In addition, information about other relevant analgesic preoperative or intraoperative medications will be gathered. Other potentially confounding intraoperative factors such as vasopressor use/amount, fluids or blood administered, total anesthesia time, etc. will be recorded. Among this group of breast surgeons, there is relative homogeneity in anatomical technique and tissue disturbance, although there is some variation in dissection technique. Detailed assessment of surgical technique will include primary surgeon, duration of surgery, presence of bilateral surgery, type of surgery (total mastectomy, segmental mastectomy), performance of nodal dissection (axillary or sentinel node), mass of breast tissue excised, length of incision, predominant mode of dissection, nerve handling, and presence and type of reconstruction.

Perioperative acute pain assessment: Initial pain score upon arrival will be assessed by PACU nursing staff and/or anesthetist. One hour after PACU arrival, patient will be assessed by research study personnel, being asked to rate pain at rest, with arm movement, and with maximal deep inspiration using the pain verbal rating scale (VRS). The Perioperative Pain Service, which is comprised of acute pain specialists, anesthesia residents, and a nurse practitioner, rounds on postoperative patients on Post-op Day (POD) 0 and 1. Accordingly, pain scores at rest, with arm movement and with deep inspiration at these two timepoints will be assessed. In addition, opioid consumption and adjuvant analgesic use will be assessed. Upon discharge, which is typically on POD1 or 2, total postoperative opioid use/hours of postoperative time as inpatient will be calculated and expressed in morphine equivalent units/hr. On postoperative day 1, patients will undergo brief bedside QST (as at preoperative evaluation, described above), PCS, and Coping Strategies Questionnaire.

Postoperative follow-up and assessment of subacute and persistent pain, changes in psychosocial and psychophysical functioning: Follow up assessments will be made at 2 weeks, 3 mo, 6 mo, and 1 year. Patients are seen by the primary surgeon or nurse practitioner, as well as by collaborator Ann Partridge and other oncologists at these times. In collaboration with these practitioners, we will assess patients' degree of persistent pain using the BCPQ, BPI and VRS. Additionally, the brief QST and psychosocial questionnaires will be re-administered at 6 months and 1 year postoperatively.

Collection of sample for future genetic testing: In order to obtain genetic information about particular sites of variability that may impact post-surgical pain, we will collect saliva samples from using the Oragene Self-Collection kit. This procedure is non-invasive, safe, effective, and widely used.

Statistical analysis: The primary outcome measure will be the calculated Pain Burden Index (PBI) at 1 year post-mastectomy. The PBI at one year post-mastectomy will be tested for significant associations with potentially predictive preoperatively assessed variables (psychophysical (QST), psychosocial, demographic, functional, medical and surgical variables) using t-tests for categorical predictors and linear regression for continuous predictors. Results of all tests will be summarized with descriptive statistics and both unadjusted p-values and p-values adjusted using Holm's procedure to control the family-wise error rate. In terms of data management and analysis, attention will be paid to identification of multi-colinearity among covariates, and redundant factors may be eliminated from further multivariable analyses.

Power analysis: Using our cross sectional data, in which roughly 35% of patients experienced persistent post-mastectomy pain beyond 1 year after mastectomy, a calculated effect size between pain and no pain groups for each of the psychosocial and psychophysical variables was determined. Effect sizes, which we assume will be similar in the proposed study, ranged from 0.06 to 0.70. With 200 patients we will have 80% power at a two-sided alpha level of 0.05 to detect effect sizes of 0.40 or greater, which were observed in 7 of the variables considered. Further corroborating the feasibility of adequate power with a sample size of 200, several smaller studies have also detected differences in QST between patients with and without chronic postsurgical pain after thoracotomy, shoulder surgery, and surgery to correct chest wall deformation.

ELIGIBILITY:
Inclusion criteria:

1. Female
2. Aged 18-80 years
3. Scheduled for total or partial mastectomy
4. Willingness to undergo psychophysical and psychosocial testing
5. Willingness to participate in long-term follow-up

Exclusion criteria:

1. Scheduled for biopsy only
2. Pregnant

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing partial or total mastectomy
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2014-10; Primary Completion 2017-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Persistent mastectomy pain | 1 year
  based the breast cancer pain questionnaire, which assesses multiple related body areas, severity and frequency of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zinboonyahgoon N, Vlassakov K, Lirk P, Spivey T, King T, Dominici L, Golshan M, Strichartz G, Edwards R, Schreiber K. Benefit of regional anaesthesia on postoperative pain following mastectomy: the influence of catastrophising. Br J Anaesth. 2019 Aug;123(2):e293-e302. doi: 10.1016/j.bja.2019.01.041. Epub 2019 Mar 28. PMID 31331591
- [Derived] Schreiber KL, Zinboonyahgoon N, Xu X, Spivey T, King T, Dominici L, Partridge A, Golshan M, Strichartz G, Edwards RR. Preoperative Psychosocial and Psychophysical Phenotypes as Predictors of Acute Pain Outcomes After Breast Surgery. J Pain. 2019 May;20(5):540-556. doi: 10.1016/j.jpain.2018.11.004. Epub 2018 Nov 23. PMID 30476655